CLINICAL TRIAL: NCT07325786
Title: A Novel Method for the Examination of Infected Wound Specimens: Percutaneous Wound Sampling With Analysis in Blood Culture (PERKA-B) Method
Brief Title: Percutaneous Wound Sampling With Analysis in Blood Culture (PERKA-B) Method
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Bülent M. Ertuğrul (Other)
Collaborators: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Dr. Bülent M. Ertuğrul, Prof. Dr., Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ADU-PERKAB-WOUND
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Wound Infection Bacterial; Identification
Keywords: Wound infection; Causative bacteria; Culture method
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Intervention Model Description: Percutaneous Wound Sampling with Analysis in Blood Culture (PERKA-B) Method:
  Tissue samples were homogenized in 5 mL of sterile saline and vortexed at 2800-3000 rpm for 2 minutes. An aliquot was collected for standard culture, after which the remaining suspension was aseptically aspirated using a 5 mL sterile syringe and inoculated into a blood culture bottle. The inoculated bottles were incubated in an automated blood culture system, and growth signals were continuously monitored. The maximum incubation period was set at 5 days; samples with no growth signal at the end of this period were considered negative.
  Upon detection of microbial growth, a sample from the blood culture bottle was subcultured onto 5% sheep blood agar and MacConkey agar plates and incubated aerobically at 35°C. Culture plates were examined for microbial growth at 24 hours. If no growth was observed, incubation was continued and plates were re-examined at 48 hours post-inoculation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Wound Sampling with Analysis in Blood Culture (PERKA-B) Method (Experimental): Percutaneous Wound Sampling with Analysis in Blood Culture (PERKA-B) Method:
  Tissue samples were homogenized in 5 mL of sterile saline and vortexed at 2800-3000 rpm for 2 minutes. An aliquot was collected for standard culture, after which the remaining suspension was aseptically aspirated using a 5 mL sterile syringe and inoculated into a blood culture bottle. The inoculated bottles were incubated in an automated blood culture system, and growth signals were continuously monitored. The maximum incubation period was set at 5 days; samples with no growth signal at the end of this period were considered negative.
  Upon detection of microbial growth, a sample from the blood culture bottle was subcultured onto 5% sheep blood agar and MacConkey agar plates and incubated aerobically at 35°C. Culture plates were examined for microbial growth at 24 hours. If no growth was observed, incubation was continued and plates were re-examined at 48 hours post-inoculation.
  Interventions: Procedure: Tissue culture collection
- Standart Microbiological analyses (Experimental): Five milliliters (mL) of sterile saline were added to the sterile tube containing the tissue specimen. The tube was mixed for 2 minutes using a vortex mixer set at 2800-3000 revolutions per minute (rpm).
  From the resulting fluid suspension, 0.05 mL was inoculated onto 5% sheep blood agar and MacConkey agar using a sterile loop under aseptic conditions. The inoculated 5% sheep blood agar and MacConkey agar plates were incubated at 35°C. 5% sheep blood agar and MacConkey agar'a inocule edilen Culture plates were examined for microbial growth at 24 hours. If no growth was observed, the plates were re-incubated and re-evaluated at 48 hours after inoculation.
  Interventions: Procedure: Tissue culture collection

INTERVENTIONS:
Procedure: Tissue culture collection — After removal of necrotic tissue under sterile conditions, an adequate tissue specimen was obtained from the infected area using surgical techniques and placed into a sterile plain tube.

SUMMARY:
The aim of this study was to evaluate whether there is a difference in pathogen detection rates when tissue samples obtained from infected wound sites are processed using standard microbiological methods compared with inoculation into blood culture bottles using a predefined protocol.

DETAILED DESCRIPTION:
Wound infections represent a major global public health problem from clinical, epidemiological, and economic perspectives. Although the incidence of surgical site infections varies by region, the global rate is estimated to be approximately 2-3% . Chronic wounds, such as diabetic foot ulcers, venous ulcers, and pressure ulcers, constitute a similarly significant burden, with their prevalence increasing steadily worldwide. Recent estimates indicate that global expenditures related to wounds and wound infections have reached 148 billion US dollars. A substantial proportion of these costs is attributable to prolonged hospitalizations and antibiotic therapy.

Rational antibiotic use in wound infections relies primarily on the identification of the causative pathogen and determination of its antimicrobial susceptibility profile through microbiological examination of appropriate clinical specimens. Because superficially collected samples carry a high risk of contamination, deep tissue biopsy or aspirate specimens are generally considered more reliable than swab samples. In routine clinical microbiology practice, standard examination of wound specimens involves inoculation onto 5% sheep blood agar in combination with MacConkey or eosin methylene blue (EMB) agar. These media are incubated at 35°C for 24 hours and subsequently evaluated. If no growth is observed, incubation is extended for an additional 24 hours, and cultures without growth after 48 hours are reported as negative. When growth is detected, further identification of the isolates is performed.

Despite meticulous specimen collection, a substantial proportion of wound samples continue to yield negative culture results. Previous investigations have documented culture-negative rates of approximately 12% in diabetic foot infections, 19% in chronic wound infections, and 10-15% in surgical site infections. In such circumstances, clinicians are often obliged to initiate empirical antimicrobial therapy when microbiological analyses fail to identify a causative pathogen, despite strong clinical evidence of infection. This approach may lead to unwarranted antibiotic administration or reliance on broad-spectrum agents, thereby increasing the risk of adverse patient outcomes and contributing to elevated healthcare expenditures. Consequently, refinement of microbiological diagnostic techniques is imperative to ensure accurate pathogen identification and to facilitate the rational selection of antimicrobial therapy.

Media used in automated blood culture systems are enriched compared with conventional solid media, such as 5% sheep blood agar, MacConkey agar, and EMB agar, and are specifically designed to enhance microbial recovery. In addition, the longer incubation periods used in these systems may further improve pathogen detection. Although blood culture systems are routinely used to detect microorganisms in blood samples obtained from peripheral veins of patients with suspected bloodstream infections, there is currently no standardized protocol for the inoculation of non-blood clinical specimens into blood culture bottles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with infected wounds

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Conventional culture vs PERKA-B Method | 3 months
  In this study, diagnostic performance measures will be calculated to evaluate the classification performance of blood culture relative to conventional culture in terms of positive and negative results.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Department of Plastic, Reconstructive and Aesthetic Surgery, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Microbiological data from tissue samples taken from infected wound of patients will be shared.
Supporting Information: CSR
Time Frame: Start date: February 1, 2026 End date: April 1, 2026
Access Criteria: Personal data and supporting information will be shared via a website accessible to researchers involved in the study. Only microbiological results of tissue samples will be available there.
URL: https://www.gedaclinic.com/

REFERENCES:
- [Background] Swanson T, Ousey K, Haesler E, Bjarnsholt T, Carville K, Idensohn P, Kalan L, Keast DH, Larsen D, Percival S, Schultz G, Sussman G, Waters N, Weir D. IWII Wound Infection in Clinical Practice consensus document: 2022 update. J Wound Care. 2022 Dec 1;31(Sup12):S10-S21. doi: 10.12968/jowc.2022.31.Sup12.S10. PMID 36475844
- [Background] Senneville E, Albalawi Z, van Asten SA, Abbas ZG, Allison G, Aragon-Sanchez J, Embil JM, Lavery LA, Alhasan M, Oz O, Uckay I, Urbancic-Rovan V, Xu ZR, Peters EJG. IWGDF/IDSA guidelines on the diagnosis and treatment of diabetes-related foot infections (IWGDF/IDSA 2023). Diabetes Metab Res Rev. 2024 Mar;40(3):e3687. doi: 10.1002/dmrr.3687. Epub 2023 Oct 1. PMID 37779323
- [Background] Rondas AA, Halfens RJ, Schols JM, Thiesen KP, Trienekens TA, Stobberingh EE. Is a wound swab for microbiological analysis supportive in the clinical assessment of infection of a chronic wound? Future Microbiol. 2015;10(11):1815-24. doi: 10.2217/fmb.15.97. PMID 26597427
- [Background] Krukerink M, Kievit J, Marang-van de Mheen PJ. Evaluation of routinely reported surgical site infections against microbiological culture results: a tool to identify patient groups where diagnosis and treatment may be improved. BMC Infect Dis. 2009 Nov 10;9:176. doi: 10.1186/1471-2334-9-176. PMID 19900294
- [Background] Macdonald KE, Boeckh S, Stacey HJ, Jones JD. The microbiology of diabetic foot infections: a meta-analysis. BMC Infect Dis. 2021 Aug 9;21(1):770. doi: 10.1186/s12879-021-06516-7. PMID 34372789
- [Background] Stevens DL, Bisno AL, Chambers HF, Dellinger EP, Goldstein EJ, Gorbach SL, Hirschmann JV, Kaplan SL, Montoya JG, Wade JC; Infectious Diseases Society of America. Practice guidelines for the diagnosis and management of skin and soft tissue infections: 2014 update by the Infectious Diseases Society of America. Clin Infect Dis. 2014 Jul 15;59(2):e10-52. doi: 10.1093/cid/ciu444. PMID 24973422
- [Background] Ertugrul B, Uckay I, Schoni M, Peter-Riesch B, Lipsky BA. Management of diabetic foot infections in the light of recent literature and new international guidelines. Expert Rev Anti Infect Ther. 2020 Apr;18(4):293-305. doi: 10.1080/14787210.2020.1730177. Epub 2020 Feb 19. PMID 32052672
- [Background] Sen CK. Human Wound and Its Burden: Updated 2025 Compendium of Estimates. Adv Wound Care (New Rochelle). 2025 Sep;14(9):429-438. doi: 10.1177/21621918251359554. Epub 2025 Jul 14. PMID 40660772
- [Background] Mengistu DA, Alemu A, Abdukadir AA, Mohammed Husen A, Ahmed F, Mohammed B, Musa I. Global Incidence of Surgical Site Infection Among Patients: Systematic Review and Meta-Analysis. Inquiry. 2023 Jan-Dec;60:469580231162549. doi: 10.1177/00469580231162549. PMID 36964747